CLINICAL TRIAL: NCT00135109
Title: A Multi-Center, Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Trial to Assess the Efficacy and Safety of SPM 927 (200, 400, and 600mg/Day) in Subjects With Painful Distal Diabetic Neuropathy
Brief Title: Trial to Assess the Efficacy and Safety of SPM 927 (200, 400, and 600mg/Day) in Subjects With Painful Distal Diabetic Neuropathy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: UCB Pharma (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SP0768
Record Dates: First submitted 2005-08-23; First posted 2005-08-25 (Estimated); Last update posted 2014-09-22 (Estimated); Status verified 2010-02

CONDITIONS: Diabetic Neuropathies
MeSH Terms: conditions — Diabetic Neuropathies | interventions — 2-(acetylamino)-3-methoxy-N-(phenylmethyl)-, (2R)-

INTERVENTIONS:
Drug: SPM 927

SUMMARY:
This phase 3 trial is being conducted at approximately 80 sites in the United States (U.S.) to investigate whether lacosamide (SPM 927) at different doses reduces pain in subjects with diabetic neuropathy. Approximately 455 subjects will be randomized to placebo or to one of three doses of lacosamide. To qualify for this trial, subjects with symptoms of painful distal diabetic neuropathy ranging in duration from 6 months to 5 years must have an average pain intensity of greater than or equal to 4 on an 11-point Likert scale (0-10 scale) during the 7 day period prior to the start of treatment.

To determine what effect lacosamide has on diabetic neuropathic pain, subjects will use a diary to record their daily pain intensity (morning and evening; and pain interference with sleep (morning) and activity (evening). Use of rescue medication (acetaminophen) and subjects' quality of life will be investigated. In addition, the safety and tolerability of the different doses of lacosamide will be investigated.

ELIGIBILITY:
Inclusion Criteria:

* Diabetic neuropathy

Exclusion Criteria:

* Subject has previously participated in this trial or subject has previously been assigned to treatment in a trial of the drug under investigation in this trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 654 (Actual)
Dates: Start 2004-10; Primary Completion 2005-12 (Actual); Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
To investigate the efficacy of 200, 400, and 600mg/day of lacosamide compared with placebo in reducing pain in subjects with painful distal diabetic neuropathy.

SECONDARY OUTCOMES:
To investigate the effect of lacosamide on subjects' perception of pain, sleep, activity, and quality of life, as well as to investigate the pharmacokinetics and safety of lacosamide.

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — UCB Pharma
Locations (1):
- Schwarz, RTP, North Carolina, United States

REFERENCES:
- [Result] Shaibani A, Fares S, Selam JL, Arslanian A, Simpson J, Sen D, Bongardt S. Lacosamide in painful diabetic neuropathy: an 18-week double-blind placebo-controlled trial. J Pain. 2009 Aug;10(8):818-28. doi: 10.1016/j.jpain.2009.01.322. Epub 2009 May 5. PMID 19409861